CLINICAL TRIAL: NCT05098613
Title: Phase 1 Study of Bispecific CD19 and CD22 Chimeric Antigen Receptor Co-Expressing T Cells (CD19x22 CAR T) in Adolescent and Adult Patients With Relapsed and/or Refractory B-Non-Hodgkin's Lymphoma (B-NHL)
Brief Title: Preliminary Safety and Tolerability of CD19x22 CAR T Cells in Adolescent and Adult R/R B-NHL Patients
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-2578.cc; NCI-2021-11091 (Other: CTRP)
Record Dates: First submitted 2021-10-06; First posted 2021-10-28 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Non-Hodgkin Lymphoma; B-cell Non-Hodgkin Lymphoma (B-NHL); Mantle Cell Lymphoma (MCL); CNS Lymphoma
Keywords: Relapsed; Refractory
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, B-Cell; Lymphoma, Mantle-Cell; Recurrence

STUDY DESIGN:
Intervention Model Description: The study is a prospective single-arm Phase 1 with four dose levels. Phase 1 will determine the maximum tolerated dose of CD19x22 CAR T cells using a standard 3+3 trial design in CAR-naïve and CAR-treated patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 Relapsed/Refractory Non-CNS B-Cell Non Hodgkin Lymphoma (Experimental): Lymphodepleting chemotherapy followed by infusion of CD19x22 CAR T Cells starting at dose level 1.
  Interventions: Drug: CD19x22 CAR T Cells
- Cohort 2 Relapsed/Refractory Mantle Cell Lymphoma (Experimental): Lymphodepleting chemotherapy followed by CD19x22 CART Infusion starting at dose level 2.
  Interventions: Drug: CD19x22 CAR T Cells
- Cohort 3: Relapsed and/or Refractory Primary CNS Lymphoma OR secondary CNS Lymphoma (Experimental): Lymphodepleting chemotherapy followed by CD19x22 CAR T Infusion starting at dose level 2
  Interventions: Drug: CD19x22 CAR T Cells

INTERVENTIONS:
Drug: CD19x22 CAR T Cells — Autologous peripheral blood mononuclear cells transduced with CD19x22 CAR T lentiviral vector.

SUMMARY:
This open-label, single arm phase 1 trial aims to determine the safety and tolerability of anti-CD19 and anti-CD22 chimeric antigen receptor-expressing (CAR) T cells (CD19x22 CAR T) in adolescents and adults with relapsed/refractory (R/R) B-cell Non-Hodgkin Lymphoma (B-NHL). This trial will determine the maximum tolerated dose of CD19x22 CAR T cells using a standard 3+3 trial design.

DETAILED DESCRIPTION:
To determine the safety and tolerability of infusing CD19x22 CAR T, generated using a bicistronic vector, in adolescents and adults with R/R B-NHL, and to determine the recommended Phase II dose (RP2D).

Secondary objectives for all subjects include: 1) Feasibility of manufacturing and infusion, 2) Safety of infusion and 3) Efficacy: Descriptive characterization of complete response (CR), partial response (PR), stable disease (SD), and progressive disease (PD) at Day +90. As well, progression-free survival (PFS), overall survival (OS), duration of remission (DOR) and overall response rate (ORR) will be determined at 1 year. Efficacy will be descriptively stratified based on prior receipt of CAR-T cell therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥ 16 years of age with no upper age limit. (NOTE: the first three subjects on this trial must be ≥ 18 years of age.)

COHORT 1: Non-CNS B-NHL

1. Histologically confirmed aggressive B-cell NHL including the following types defined by World Health Organization (WHO) 2008:

   a. Diffuse Large B-Cell Lymphoma (DLBCL) not otherwise specified; T cell/histiocyte rich large B cell lymphoma; DLBCL associated with chronic inflammation; Epstein Barr Virus (EBV)+ DLBCL of the elderly; OR b. Primary mediastinal (thymic) large B cell lymphoma; OR c. Transformation to DLBCL; OR d. High grade B-cell Lymphoma (HGBL).
2. Subjects must not have any signs or symptoms of CNS disease or detectable evidence of CNS disease on magnetic resonance imaging (MRI) at screening; subjects who have been previously treated for CNS disease, but have no evidence of disease at screening are eligible for this cohort.
3. Subjects must have disease progression confirmed by either flow cytometry or immunohistochemistry (IHC), disease stabilization, or disease recurrence after at least two lines of therapy.

   a. The two lines of prior therapy must include an anthracycline and anti-CD20 monoclonal antibody treatment.

   b. Relapse or refractory after single antigen targeting CAR T cell therapy
4. Must have evaluable or measurable disease according to the revised International Working Group (IWG) Response Criteria for Malignant Lymphoma; lesions that have been previously irradiated will be considered measurable only if progression has been documented following completion of radiation therapy.

COHORT 2: MANTLE CELL LYMPHOMA (MCL)

1. Mantle Cell Lymphoma (MCL).

   a. Results of all tests conducted on the tissue at initial diagnosis and/or relapse, including, but not limited to, the MCL subtype (classic and blastoid), Ki-67 proliferation index, and TP53 mutation status should be provided if done.
2. Subjects must have relapsed and/or refractory MCL confirmed by either flow cytometry or immunohistochemistry (ICH), disease stabilization, or disease recurrence after at least two lines of therapy including any combination of the agents below:

   a. An anti-CD20-directed therapy b. A BTK inhibitor c. Anthracycline or Bendamustine d. Relapse or refractory after single antigen targeting CAR T cell therapy.
3. Must have evaluable or measurable disease according to the revised International Working Group (IWG) Response Criteria for Malignant Lymphoma; lesions that have been previously irradiated will be considered measurable only if progression has been documented following completion of radiation therapy. MCL patients without measurable nodal or extranodal disease by IWG criteria are eligible if they have bone marrow involvement of MCL at relapse

COHORT 3: PRIMARY CNS LYMPHOMA OR SECONDARY CNS LYMPHOMA

1. Subjects with relapsed and/or refractory primary CNS lymphoma (PCNSL) OR secondary CNS lymphoma (SCNSL), as defined by the following:

   a. Absence of measurable disease outside the CNS, as determined by radiographic imaging (i.e. PET/CT).

   b. Detectable CNS disease, as defined as: i. At least 1 site of measurable disease within the brain or spinal cord that is ≥ 1 cm in the longest diameter based on MRI or PET/CT imaging; OR, ii. Neoplastic B-cells detectable within the CSF or vitreous by flow cytometry or cytology.
2. Subjects must have disease progression confirmed by either flow cytometry or immunohistochemistry (IHC), disease stabilization, or disease recurrence after at least one line of therapy.

ALL COHORTS:

1. Subjects who have undergone autologous stem cell transplantation (SCT) with disease progression or relapse are eligible.
2. Subjects who have undergone allogeneic SCT will be eligible if, in addition to meeting other eligibility criteria, are:

   1. At least 100 days post-transplant,
   2. Do not have active graft versus host disease (GVHD)
3. Any standard of care systemic therapy prior to leukapheresis must follow the washout period.
4. Any steroid use (dexamethasone or prednisone) prior to apheresis must follow the washout period. Physiological replacement doses are allowable with no washout period. Topical or inhaled steroids for localized GVHD is allowable.
5. Peripheral blood CD3 count must be >0.15 x 10 (to the 6th) cells/mL within 14 days prior to proceeding with apheresis.
6. Toxicities from prior therapy must be stable and recovered to ≤ grade 1 (exceptions include non-clinically significant toxicities such as alopecia and the organ function definitions provided in inclusion criteria 12).
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2, or Karnofsky ≥ 80%.
8. Adequate organ function as defined by:

   1. Absolute neutrophil count (ANC) ≥ 500/μL
   2. Platelet count ≥ 50,000/ μL.
   3. Renal: Creatinine ≤ 2 mg/dL OR creatinine clearance (as estimated by Cockcroft Gault equation) ≥ 60 mL/min.
   4. Hepatic: Serum alanine aminotransferase (ALT)/aspartate aminotransferase (AST) ≤ 3 upper limit of normal (ULN).
   5. Total bilirubin ≤ 2 mg/dl, except in subjects with Gilbert's syndrome where a bilirubin <4.0 will be acceptable.
   6. Cardiac: Ejection fraction ≥ 40%, no evidence of physiologically significant pericardial effusion as determined by an echocardiogram (ECHO), and no clinically significant electrocardiogram (ECG) findings within 6 weeks of apheresis.
   7. Pulmonary: No clinically significant pleural effusion and;

   i. Baseline oxygen saturation must be > 92% on room air
9. Females of childbearing potential must have a negative serum pregnancy test (females who have undergone surgical sterilization or who have been postmenopausal for at least 6 months are not considered to be of childbearing potential).
10. Subjects of childbearing or child-fathering potential must be willing to practice birth control from the time of enrollment on this study and for 12 months after receiving the CD19x22 infusion; females of childbearing potential must have a negative pregnancy test.

21. Must be able to give informed consent; subjects unable to give informed consent will not be eligible for this study.

22. Be able to consent to long-term follow-up protocol (#20-0188).

Exclusion Criteria:

1. Age < 16 years of age.
2. Patient who is intolerant of contrast-enhanced MRI due to allergic reactions to contrast agents. Only applicable to Cohort 3.
3. History of other malignancies, unless they have been disease free for at least 3 years. Exceptions include non-melanoma skin cancer or carcinoma in situ and localized prostate cancer not on active treatment.
4. Uncontrolled fungal, bacterial, viral, or other infection requiring antimicrobials for management; uncomplicated infections are permitted if responding to active treatment.
5. Known history of infection with human immunodeficiency virus (HIV) or hepatitis B (hepatitis B surface antigen [HBsAg] positive) or hepatitis C.
6. History of known myocardial infarction, cardiac angioplasty or stenting, unstable angina, or other clinically significant cardiac disease within 12 months of enrollment or have cardiac atrial or cardiac ventricular lymphoma involvement.
7. Venous thrombosis or embolism not managed on a stable regimen of anticoagulation.
8. Any medical condition that in the judgement of the sponsor is likely to interfere with assessment of safety or efficacy of study treatment.
9. History of severe immediate hypersensitivity reaction to any of the agents used in this study.
10. Pregnancy (serum pregnancy test must be obtained at time of enrollment for females of childbearing potential and to be repeated 72 hours prior to lymphodepleting chemotherapy regimen); females who have undergone surgical sterilization or who have been postmenopausal for at least 6 months are not considered to be childbearing potential.
11. Lactating.
12. In the investigator's judgment, the subject is unlikely to complete all protocol required study visits or procedures, including follow up visits, or comply with the study requirements for participation.
13. Unwilling to participate in long-term follow-up protocol that is required if CAR T cell therapy is administered at CU Anschutz.

LYMPHODEPLETING CHEMOTHERAPY ELIGIILITY:

In order to proceed with lymphodepleting chemotherapy, enrolled participants must meet all eligibility criteria below within 72 hours prior to lymphodepletion, unless otherwise specified:

* If the participant received bridging therapy after apheresis, confirmation of disease reevaluation is required. It must be within 6 weeks of initiation of LD chemotherapy.

  * Confirmation that the participant has met the washout period for bridging therapy.
* Negative serum pregnancy test (for women of childbearing potential)
* Adequate organ function as defined by:

  * Absolute neutrophil count (ANC) ≥ 500/μL.
  * Platelet count ≥ 50,000/ μL.
  * Renal: Creatinine ≤ 2 mg/dL OR creatinine clearance (as estimated by Cockcroft Gault equation) ≥ 60 mL/min.
  * Hepatic: Serum alanine aminotransferase (ALT)/aspartate aminotransferase (AST) ≤ 3 upper limit of normal (ULN).
  * Total bilirubin ≤ 2 mg/dl, except in subjects with Gilbert's syndrome where a bilirubin <3.0 will be acceptable.
  * Pulmonary: No clinically significant pleural effusion and; Baseline oxygen saturation must be > 92% on room air.
  * Cardiac: Ejection fraction ≥ 45%, no evidence of physiologically significant pericardial effusion as determined by an echocardiogram (ECHO) (only if subject received bridging anthracycline or developed a significant illness prior to LD-chemo per investigator assessment.) If clinically indicated, ECHO must be performed within 2 weeks prior to LD-chemotherapy.

CD19x22 CAR T CELL INFUSION ELIGIBILITY

In order to proceed with CD19x22 CAR T Cell Infusion, enrolled participants must meet all eligibility criteria below within 24 hours prior to CD19x22 CAR T Cell infusion, unless otherwise specified:

* CD19x22 CAR T cells must have met manufacturing release criteria (unless prospectively approved by IND Sponsor, Gates Institute Medical Lead, and FDA).
* Confirmation that the site has Anakinra and Ruxolitinib in stock and available (should IEC-HS treatment be required).
* ECOG ≤2 or Karnofsky≥ 50%.
* Clinically stable without evidence of vital sign instability, including the lack of supportive vasoactive drugs or intensive care unit support.
* Oxygen saturation > 92% on room air; cannot be on supplemental oxygen.
* No evidence of uncontrolled, significant tumor lysis syndrome prior to cell infusion per investigator assessment.
* No evidence of rapidly progressive NHL per investigator determination.
* Participants' temperature is <38.0 °C within 48 hours prior to cell infusion. (If the source of fever cannot be identified [after thorough infectious disease work-up], and the suspected cause is underlying malignancy, discussion and approval by the Gates Institute Medical Lead may allow continued infusion of CD19x22 cells. This should be appropriately documented in the patient's medical record.
* Liver transaminase (ALT and AST) < 5 x institutional ULN (< grade 3) based on age- and laboratory- specific normal ranges.
* Adequate renal function as defined by creatinine ≤ 2 mg/dL OR creatinine clearance (as estimated by the Cockcroft- Gault equation) ≥ 60 mL/min.

If these criteria are not met, measures can be taken to resolve the underlying condition(s). If successful, cells may be infused up to (and including) 7 days following the time of the planned infusion with no additional lymphodepletion. If the CD19x22 CAR T Cell infusion is delayed more than 7 days, lymphodepleting chemotherapy MAY be repeated, per the investigator's discretion. Prior to commencing a second round of lymphodepletion, participants must meet lymphodepletion criteria described above.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2021-12-21 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Overall safety and tolerability of CD19x22 CAR T Therapy in CAR-naive and CAR-treated subjects | 12 Months Post Infusion
  Assessed by Type, Frequency, and Severity of Adverse Events (AEs). All AEs, including laboratory abnormalities, will be graded using the National Cancer Institute's (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 grading criteria.
Determine the Recommended Phase II Dose (RP2D) Level | 30 Days Post Infusion
  Incidence and frequency of Grade 3-5 toxicity occurring within the dose limiting toxicity (DLT) period post CD19x22 CAR T infusion. Grades 3-5 adverse events (AEs) are defined as Severe, Life-Threatening, and Fatal.

SECONDARY OUTCOMES:
Feasibility of Manufacturing CD19x22 CAR T | Day 0 (Infusion)
  The feasibility of manufacturing the desired dose of anti-CD19x22 CAR T cells will be established using the percentage of patients for whom the desired dose of CAR T cells was successfully produced.
Evaluate Safety of Infusion | 30 Days Post Infusion
  Percentage of study participants who receive CD19x22 CAR T infusion without infusion reaction
Evaluate Clinical Efficacy of CD19x22 CAR T | 12 Months Post Infusion
  Clinical efficacy is defined through Lugano response criteria at Day +60 (Cohort 2 only), Day +90, 6 months, and 1 year. Efficacy will be stratified based on prior receipt of CAR T cell therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Manali Kamdar, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No